CLINICAL TRIAL: NCT02350816
Title: An Open-Label Extension of Study HGT-SAN-093 Evaluating the Safety and Efficacy Study of HGT-1410 (Recombinant Human Heparan N Sulfatase) Administration Via an Intrathecal Drug Delivery Device in Pediatric Patients With Mucopolysaccharidosis Type IIIA Disease
Brief Title: An Extension Study to Determine Safety and Efficacy for Pediatric Patients With MPS Type IIIA Disease Who Participated in Study HGT-SAN-093.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Completion of follow-up period
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP610-201; 2014-003960-20 (EudraCT Number)
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Sanfilippo Syndrome; Mucopolysaccharidosis (MPS)
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HGT-1410 Q2W in Study HGT-SAN-093 randomized to HGT-1410 Q2W (Active Comparator): Patients in Group 1 will continue HGT-1410 treatment at a dose of 45 mg administered every 2 weeks (Q2W) starting at Week 50, with a cumulative treatment period of up to 42 months (168 weeks) . HGT-1410 will be administered intrathecally (IT) by an indwelling intrathecal drug delivery device (IDDD).
  HGT-SAN-093 = NCT02060526
  Interventions: Drug: HGT-1410
- HGT-1410 Q4W in Study HGT-SAN-093 randomized to HGT-1410 Q4W (Active Comparator): Patients in Group 2 will continue HGT-1410 treatment at a dose of 45 mg administered every 4 weeks (Q4W) starting at Week 52, with a cumulative treatment period of up to 42 months (168 weeks). HGT-1410 will be administered intrathecally (IT) by an indwelling intrathecal drug delivery device (IDDD).
  Interventions: Drug: HGT-1410
- no-treatment in Study HGT-SAN-093 randomized to HGT-1410 Q2W (Active Comparator): Patients in Group 3A will receive an IDDD following informed consent and will be randomized in a 1:1 allocation ratio to begin HGT-1410 treatment at a dose of 45 mg administered every 2 weeks (Q2W) starting at Week 0 of the extension study, with a cumulative treatment period of up to 30 months (120 weeks). HGT-1410 will be administered intrathecally (IT) by an indwelling intrathecal drug delivery device (IDDD).
  Interventions: Drug: HGT-1410
- no-treatment in Study HGT-SAN-093 randomized to HGT-1410 Q4W (Active Comparator): Patients in Group 3B will receive an IDDD following informed consent and will be randomized in a 1:1 allocation ratio to begin HGT-1410 treatment at a dose of 45 mg administered every 4 weeks (Q4W) starting at Week 0 of the extension study, with a cumulative treatment period of up to 30 months (120 weeks). HGT-1410 will be administered intrathecally (IT) by an indwelling intrathecal drug delivery device (IDDD).
  Interventions: Drug: HGT-1410

INTERVENTIONS:
Drug: HGT-1410 — HGT-1410 administered according to Patient Group assignment.
  Other Names: Recombinant Human Heparan N Sulfatase

SUMMARY:
This extension study will allow participants to continue receiving treatment with HGT-1410 and to initiate treatment in patients who received no-treatment in Study HGT-SAN-093, and will evaluate the long-term safety and efficacy of the study drug.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be considered eligible for enrollment:

1. Patient has completed through at least the Week 48 visit of Study HGT-SAN-093
2. The patient's parent(s) or legally authorized guardian(s) must have voluntarily signed an Institutional Review Board- (IRB-)/ Independent Ethics Committee- (IEC-) approved informed consent form after all relevant aspects of the study have been explained and discussed. Consent of the patient's parent(s) or legally authorized guardian(s) and the patient's assent, as relevant, must be obtained

Exclusion Criteria:

Patients will be excluded from the study if any of the following criteria are met:

1. The patient, if randomized to treatment in Study HGT-SAN-093, has experienced a decline of more than 20 points in the BSID-III cognitive DQ score between Baseline and the Week 48 visit in Study HGT-SAN-093, AND, upon individual evaluation by the Investigator, has been deemed a treatment failure*
2. The patient has experienced, in the opinion of the Investigator, a safety or medical issue that contraindicates treatment with HGT-1410, including but not limited to clinically relevant intracranial hypertension, severe infusion-related reactions after treatment with HGT-1410, uncontrollable seizure disorder
3. The patient has a known hypersensitivity to any of the components of HGT-1410
4. The patient is enrolled in another clinical study, other than HGT-SAN-093, that involves clinical investigations or use of any investigational product (drug or [intrathecal/spinal] device) within 30 days prior to study enrollment or at any time during the study
5. The patient has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to airway compromise or other conditions
6. The patient has a condition that is contraindicated as described in the SOPH-A-PORT® Mini S IDDD Instructions for Use, including:

   1. The patient has had, or may have, an allergic reaction to the materials of construction of the SOPH-A-PORT ® Mini S device
   2. The patient's body size is too small to support the size of the SOPH-A-PORT ® Mini S Access Port, as judged by the Investigator
   3. The patient's drug therapy requires substances known to be incompatible with the materials of construction
   4. The patient has a known or suspected local or general infection
   5. The patient is at risk of abnormal bleeding due to a medical condition or therapy
   6. The patient has one or more spinal abnormalities that could complicate safe implantation or fixation
   7. The patient has a functioning CSF shunt device
   8. The patient has shown an intolerance to an implanted device
7. The patient is unable to comply with the protocol (eg, is unable to return for safety evaluations, or is otherwise unlikely to complete the study) as determined by the Investigator

   * All treated patients in Study HGT-SAN-093 will have their cognitive development assessed at the Week 48 Visit in Study HGT-SAN-093. If a decline from Baseline of 20 points or less in the BSID-III DQ score is observed, then the patient may proceed into the Study SHP-610-201 without further evaluation. If a decline from Baseline of more than 20 points in DQ score is observed, then an individual evaluation by the Investigator will occur to determine if the patient is a treatment failure. This individual evaluation will take into account the DQ scores, VABS-II score, physical status, and any other information available for that patient at that time. If the Investigator deems the patient to be a treatment failure, then the patient may not enter the Study SHP-610-201

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Chu Bicetre, Le Kremlin-Bicêtre, Paris, France
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany
- Azienda Socio Sanitaria Territoriale - Asst di Monza, Monza, Italy
- Academisch Medisch Centrum Amsterdam, Amsterdam, Netherlands
- Hospital Universitario Vall D'hebron - Ppds, Barcelona, Spain
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant enrolled in the study on 08 April 2015 and last participant last follow-up on 12 April 2019.
Pre-assignment Details: A total of 17 participants were enrolled and completed treatment period in the study.
Groups:
- Group 1: Participants continued HGT-1410 treatment from HGT-SAN-093 (NCT02350816) study at a dose of 45 milligrams (mg) administered intrathecally (IT) via IT drug delivery device (IDDD) every 2 weeks (Q2W) started at Week 50, with a cumulative treatment period of up to 42 months (168 weeks).
- Group 2: Participants continued HGT-1410 treatment from HGT-SAN-093 (NCT02350816) study at a dose of 45 mg administered intrathecally IDDD every 4 weeks (Q4W) started at Week 52, with a cumulative treatment period of up to 42 months (168 weeks).
- Group 3A: Participants in Group 3A were not treated in HGT-SAN-093 (NCT02350816) study. Participants received HGT-1410 treatment at a dose of 45mg administered intrathecally IDDD Q2W started at Week 0 of the current extension study (SHP610-201=2014-003960-20), with a cumulative treatment period of up to 30 months (120 weeks).
- Group 3B: Participants in Group 3B were not treated in HGT-SAN-093 (NCT02350816) study. Participants received HGT-1410 treatment at a dose of 45mg administered intrathecally via IDDD Q4W started at Week 0 of the current extension study (SHP610-201=2014-003960-20), with a cumulative treatment period of up to 30 months (120 weeks).
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Started | 7 | 6 | 2 | 2
Completed (Participants who completed treatment period.) | 7 | 6 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who had the IDDD implant or received at least 1 dose of investigational product in the extension study (SHP610-201 [NCT02350816]).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B | Total
Number analyzed (Participants) | 7 | 6 | 2 | 2 | 17
Age, Continuous [Mean (Standard Deviation); unit: Months] | 29.64 (9.989) | 31.62 (8.598) | 40.40 (5.798) | 36.95 (7.142) | 32.47 (8.941)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 0 | 10
  Male | 2 | 3 | 0 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 5 | 2 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 6 | 2 | 2 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Based on Type, Severity and Relationship to Treatment Drug
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered as a pharmaceutical product that did not necessarily have a causal relationship with this treatment. TEAEs was defined as all AEs from the time of initial IDDD implantation (or first dose if earlier) in either Study NCT02060526 (HGT-SAN-093) or Study NCT02350816 (SHP-610-210) to the data cutoff date (28 Jun 2017), or 30 days after the date of the last dose or 2 weeks after the date of device explant (whichever was later) if early termination occurred. Treatment-emergent AEs were summarized by type (serious, life-threatening), severity (mild, moderate, severe) and degree of relationship to investigational product (Intrathecal Drug Delivery Device (IDDD), device surgical procedure, or intraThecal administration of HGT-1410).
Time Frame: From start of study drug administration up to follow-up (Week 276)
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 7 | 6 | 2 | 2
Participants
  Participants with TEAEs | 7 | 6 | 2 | 2
  Participants with Serious TEAEs | 6 | 6 | 0 | 1
  Participants with Life-Threatening TEAEs | 0 | 0 | 0 | 0
  Participants with Mild TEAEs | 0 | 0 | 1 | 1
  Participants with Moderate TEAEs | 4 | 4 | 1 | 1
  Participants with Severe TEAEs | 3 | 2 | 9 | 9
  Participants with HGT-1410 Related TEAEs | 5 | 5 | 1 | 1
  Participants with Surgery Related TEAEs | 6 | 6 | 1 | 1
  Participants with IDDD Related TEAEs | 5 | 6 | 0 | 1
  Participants with IT Administration Related TEAEs | 3 | 6 | 0 | 1

2. Primary Outcome: Number of Participants With Positive Anti-Recombinant Human Heparan N-Sulfatase (rhHNS) Antibody Status in Serum
Description: Number of participants with positive anti-rhHNS antibody status in serum were reported.
Time Frame: Up to 120 weeks
Population: Safety population consisted of all participants who had the IDDD implant or received at least 1 dose of investigational product in the extension study (SHP610-201 [NCT02350816]). The last observed time point data was presented for outcome measure data.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 7 | 6 | 2 | 2
Participants | 7 | 6 | 2 | 2

3. Primary Outcome: Area Under Curve (AUC) of Recombinant Human Heparan N-Sulfatase (rhHNS) Concentration in Cerebro Spinal Fluid (CSF)
Description: No sufficient pharmacokinetic (PK) samples were collected and analyzed due to early termination of the study.
Time Frame: Week 0 and 48
Population: No sufficient PK samples were collected and analyzed due to early termination of the study.
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Primary Outcome: Area Under Curve (AUC) of Recombinant Human Heparan N-Sulfatase (rhHNS) Concentration in Serum
Description: No sufficient PK samples were collected and analyzed due to early termination of the study.
Time Frame: Week 0, 48 and 96
Population: No sufficient pharmacokinetic (PK) samples were collected and analyzed due to early termination of the study.
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Levels of Glycosaminoglycan (GAG) Concentration in Cerebro Spinal Fluid (CSF)
Description: Levels of GAG concentration in CSF was reported. Last measurable data was presented for respective participant up to their last observed time point.
Time Frame: Up to Week 120
Population: Safety population consisted of all participants who had the IDDD implant or received at least 1 dose of investigational product in the extension study (SHP610-201 [NCT02350816]). Here the number of participants analyzed signifies participants who were evaluable for this measure at specific category.
Measure: Number; unit: micromoles (μmol)
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 7 | 6 | 2 | 2
micromoles (μmol)
  Participant 1: Week 16: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1: Week 16 |  |  |  | 3.67
  Participant 2: Week 60: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2: Week 60 |  | 1.52 |  |
  Participant 3: Week 86: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3: Week 86 | 0.698 |  |  |
  Participant 4: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 4: Week 72 |  | 1.5 |  |
  Participant 5: Week 44: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 5: Week 44 |  |  | 0.592 |
  Participant 6: Week 72: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 6: Week 72 | 2.62 |  |  |
  Participant 7: Week 120: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 7: Week 120 |  | 1.26 |  |
  Participant 8: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 8: Week 72 |  | 2.49 |  |
  Participant 9: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 9: Week 72 |  | 1.77 |  |
  Participant 10: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 10: Week 72 |  | 2.13 |  |
  Participant 11: Week 60: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 11: Week 60 | 1.35 |  |  |
  Participant 12: Week 96: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 12: Week 96 | 0.491 |  |  |
  Participant 13: Week 84: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 13: Week 84 | 2.84 |  |  |
  Participant 14: Week 62: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 14: Week 62 | 4.05 |  |  |
  Participant 15: Week 60: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 15: Week 60 | 1.63 |  |  |
  Participant 16: Week 20: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 16: Week 20 |  |  | 0.699 |
  Participant 17: Week 8: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 17: Week 8 |  |  |  | 2.59

6. Primary Outcome: Levels of Glycosaminoglycan (GAG) Concentration in Urine
Description: Levels of GAG concentration in Urine were reported. Last measurable data was presented for respective participant up to their last available time point.
Time Frame: Up to Week 120
Population: as for outcome 5
Measure: Number; unit: percentage of GAG
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 7 | 6 | 2 | 2
percentage of GAG
  Participant 1: Week 16: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 1: Week 16 |  |  |  | 48.562684655
  Participant 2: Week 60: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 2: Week 60 |  | 36.6 |  |
  Participant 3: Week 86: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 3: Week 86 | 23.814294737 |  |  |
  Participant 4: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 4: Week 72 |  | 33.220498513 |  |
  Participant 5: Week 44: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 5: Week 44 |  |  | 31.266295955 |
  Participant 6: Week 72: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 6: Week 72 | 41.417183858 |  |  |
  Participant 7: Week 120: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 7: Week 120 |  | 126.08093356 |  |
  Participant 8: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 8: Week 72 |  | 41.442593994 |  |
  Participant 9: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 9: Week 72 |  | 33.736917544 |  |
  Participant 10: Week 72: number analyzed (Participants) | 0 | 1 | 0 | 0
  Participant 10: Week 72 |  | 21.063333103 |  |
  Participant 11: Week 60: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 11: Week 60 | 41.011940047 |  |  |
  Participant 12: Week 96: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 12: Week 96 | 24.508878333 |  |  |
  Participant 13: Week 84: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 13: Week 84 | 11.31179 |  |  |
  Participant 14: Week 62: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 14: Week 62 | 61.047755556 |  |  |
  Participant 15: Week 60: number analyzed (Participants) | 1 | 0 | 0 | 0
  Participant 15: Week 60 | 40.230919792 |  |  |
  Participant 16: Week 20: number analyzed (Participants) | 0 | 0 | 1 | 0
  Participant 16: Week 20 |  |  | 38.608023285 |
  Participant 17: Week 8: number analyzed (Participants) | 0 | 0 | 0 | 1
  Participant 17: Week 8 |  |  |  | 39.247789595

7. Secondary Outcome: Change From Baseline Vineland Adaptive Behavior Scales Second Edition (VABS-II)
Description: VABS-II measured adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. It was an instrument that supports the diagnosis of intellectual and developmental disabilities in participants. This test measured 5 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite ((a composite of the other four domains). Scoring was 'Usually' = 2, 'Sometimes'/Partially' = 1 or 'Never' = 0. The raw scores was converted to domain standard scores (mean 100, SD 15). Higher scores indicate undesirable behavior. Due to the premature termination of the treatment period, efficacy data were not analyzed and no efficacy conclusions were drawn.
Time Frame: Baseline, Week 120
Population: No participant was analyzed due to the premature termination of the treatment period of this study.
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in the Developmental Quotient (DQ) Assessed by Neurocognitive Tests
Description: The development quotient (DQ) was to express a neurodevelopmental/cognitive delay which was computed as a ratio and expressed as a percentage using the age equivalent score divided by the age at testing ([age-equivalent score/chronological age] × 100; range: 0, 100). Higher scores are indicative of decreased development. Neurocognitive tests included Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III), Kaufman Assessment Battery for Children, Second Edition (KABC-II), Vineland Adaptive Behavior Scales, Second Edition (VABS-II). Due to the premature termination of the treatment period, efficacy data were not analyzed and no efficacy conclusions were drawn.
Time Frame: Baseline, Week 120
Population: No participant was analyzed due to the premature termination of the treatment period of this study.
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Total Cortical Grey Matter Volume
Description: The total cortical grey matter volume was assessed by volumetric magnetic resonance imaging (MRI) of the brain. Due to the premature termination of the treatment period, efficacy data were not analyzed and no efficacy conclusions were drawn.
Time Frame: Baseline, Week 120
Population: No participant was analyzed due to the premature termination of the treatment period of this study.
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Week 276)
Arm/Group | Group 1 | Group 2 | Group 3A | Group 3B
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 6/7 | 6/6 | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=7) | Group 2 (N=6) | Group 3A (N=2) | Group 3B (N=2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Device failure (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Implant site extravasation (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=7) | Group 2 (N=6) | Group 3A (N=2) | Group 3B (N=2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (6) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (14) | 3 (4) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site extravasation (General disorders) | 1 (1) | 2 (5) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implant site swelling (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (29) | 3 (6) | 2 (12) | 2 (5)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 4 (6) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (6) | 1 (2) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (4) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 5 (11) | 1 (2) | 1 (1) | 0 (0)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stitch abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (28) | 2 (5) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 1 (3)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (6) | 0 (0) | 1 (3)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (4)
Body temperature decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
CSF protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CSF test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CSF white blood cell count increased (Investigations) | 1 (3) | 3 (4) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (6) | 0 (0) | 1 (5)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (4) | 1 (2) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Protein total increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory rate decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urine uric acid (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Demyelination (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased interest (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep terror (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated as prespecified efficacy criteria were not met and study did not yield clinical proof-of-concept, prompting a decision to discontinue further clinical development of HGT-1410. Hence efficacy parameters were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT02350816/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT02350816/SAP_001.pdf